CLINICAL TRIAL: NCT07024563
Title: A Phase 3, Open-Label, Multicenter Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Efficacy, and Safety of Ravulizumab in Pediatric Participants (2 to < 18 Years of Age) With Primary Immunoglobulin A Nephropathy (IgAN)
Brief Title: Study of Ravulizumab in Pediatric Participants With Primary IgAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D928FC00002; 2024-520167-13-00 (Other: EUCTR)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: IgAN; IgAVN; Immunoglobulin A Nephropathy; Immunoglobulin A Vasculitis Associated Nephritis; Henoch-schonlein Purpura Nephritis; IgA Vasculitis
Keywords: ravulizumab; IgAN; IgAVN; pediatric; proteinuria; glomerulonephropathy; Immunoglobulin A Nephropathy; Immunoglobulin A Vasculitis Associated Nephritis
MeSH Terms: conditions — Glomerulonephritis, IGA; IgA Vasculitis; Proteinuria | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ravulizumab (Experimental): All participants will receive a weight-based loading dose of ravulizumab on Day 1, followed by weight-based maintenance treatment with ravulizumab on Day 15 and either once every 8 weeks (q8w) thereafter or once every 4 weeks (q4w) depending on weight.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Participants will receive Ravulizumab via intravenous (IV) infusion.

SUMMARY:
The primary objectives of this study are to characterize ravulizumab pharmacokinetics (PK) and pharmacodynamics (PD), and to evaluate safety and efficacy following ravulizumab IV dosing in pediatric participants with IgAN or IgAVN.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 2 to < 18 years of age at the time of signing the informed consent or assent.
* Stable and maximum allowed or tolerated RASI (ACEI and/or ARB) dose for ≥ 3 months prior to Screening with no planned change during Screening through Week 106.
* UPCR ≥ 1.0 g/g from the mean of 3 first morning voids (FMV) collected within 1 week during the Screening Period
* Estimated GFR ≥ 30 mL/min/1.73 m2 during Screening
* Meningococcal infection vaccine
* Haemophilus influenzae type b and Streptococcus pneumoniae vaccine
* Participants who are receiving SGLT2i, DEARA (eg, sparsentan), MRA, ERA, or GLP-1 agonists must be on a stable and maximum allowed or tolerated dose for ≥ 3 months prior to Screening with no planned change in dose through Week 34.
* Established diagnosis of primary IgAN diagnosis based on kidney biopsy within 3 years prior to Screening or during the Screening Period

Exclusion Criteria:

* Diagnosis of rapidly progressive glomerulonephritis
* Secondary forms of IgAN not in the context of primary IgAN or IgAV
* Concomitant clinically significant renal disease other than IgAN or IgAVN
* Clinical remission of IgAN/IgAVN or clinically significant improvement in proteinuria within the last 6 months.
* Uncontrolled diabetes mellitus with HbA1c > 8.5%
* History of kidney transplant or planned kidney transplant during the Primary Evaluation Period.
* History of other solid organ (heart, lung, small bowel, pancreas, or liver) or bone marrow transplant
* Splenectomy or functional asplenia
* Participants with nephrotic syndrome receiving albumin infusions or with acute kidney injury requiring dialysis within the last 6 months prior to Screening.
* Hemolytic uremic syndrome diagnosed any time prior to Screening.
* Planned urological surgery expected to influence kidney function within the study time frame.
* Congenital immunodeficiency
* Active systemic bacterial, viral, or fungal infection within 14 days prior to enrollment
* Received biologics for the treatment of IgAN or IgAVN within≤ 6 months prior to Screening

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2028-07-12 (Estimated); Study Completion 2029-11-27 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Proteinuria Based on Urine Protein to Creatinine Ratio (UPCR) at Week 34 | Baseline, Week 34

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Ravulizumab | Baseline up to Week 34
Trough Serum Concentration (Ctrough) of Ravulizumab | Baseline up to Week 34
Change From Baseline in Serum Free Complement Component 5 (C5) Concentration | Baseline up to Week 34
Change from Baseline in proteinuria based on Urine Protein to Creatinine Ratio (UPCR) at Week 10 | Baseline, Week 10
Change from Baseline in Albuminuria based on Urine Albumin to Creatinine Ratio (UACR) at Week 34 | Baseline, Week 34
Number of Participants with Partial Remission | Week 34
Annualized Total Estimated Glomerular Filtraion Rate (eGFR) over 106 weeks | Baseline up to Week 106
Change from Baseline in eGFR | Baseline, Weeks 50 and 106
Number of Participants with UPCR <0.5 gram of protein per gram of creatinine | Week 34
Number of Participants With Treatment Emergent Adverse Events, Treatment Emergent Serious Adverse Events and Adverse Events of Special Interest | Baseline up to Week 106
Number of Participants with Antidrug Antibodies to Ravulizumab and Neutralizing Antibodies | Baseline up to Week 106

CONTACTS AND LOCATIONS:
Locations (12):
- Research Site, Aurora, Colorado, United States
- China (2):
  - Research Site, Beijing
  - Research Site, Shanghai
- Italy (3):
  - Research Site, Genova
  - Research Site, Roma
  - Research Site, Torino
- Research Site, Wakayama, Japan
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Seville
- Taiwan (2):
  - Research Site, Taipei
  - Research Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR